CLINICAL TRIAL: NCT00903045
Title: Urinary Urgency Outcomes Following Propiverine Treatment for an Overactive Bladder: PRopiverine Study on Overactive Bladder Including Urgency Data (PROUD)
Brief Title: Urinary Urgency Outcomes Following Propiverine Treatment for an Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-01-08
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Propiverin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — propiverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Propiverine hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propiverine hydrochloride — Propiverine hydrochloride 20mg twice a day
  Other Names: BUP-4
  Arms: 1
Drug: Placebo — Identical placebo twice a day
  Arms: 2

SUMMARY:
Overactive bladder (OAB) is defined as "urgency, with or without urge incontinence, usually with frequency and nocturia" in the absence of local pathological or endocrine factors. Urgency is defined as "the complaint of a sudden compelling desire to pass urine that is difficult to defer" and an abnormal sensation that is distinctly different from the normal physiologic feeling of 'urge to void' that occurs during typical bladder-filling cycles.

Because up to 50% of patients with OAB experience urgency without incontinence, and because urgency is the most bothersome symptom that drives behavioral adaptations such as frequent voiding because of the very fear of urgency, this is the cornerstone symptom of OAB that indicates the diagnosis of OAB.

Even though any effective treatment for OAB must reduce the patient's sense of urgency, its subjective nature makes it difficult to measure. Therefore, the clinical efficacy of OAB treatment was traditionally measured in terms of objective surrogate parameters instead of urgency itself: for example, change in urinary frequency, incontinent episodes, number of pads and urodynamically proven detrusor overactivity, which could be measured easily and quantifiably.

Recently, several methods that measure urgency have been developed and used in clinical practice. However, the analysis questioned the clinical significance of the results; a possible reason for this being the lack of data based on urinary urgency and the use of sensitive patient-driven criteria.

Propiverine hydrochloride (1-methyl-4-piperidyl diphenylpropoxyacetate hydrochloride) is a drug with combined antimuscarinic and calcium antagonistic actions. Previous trials on the clinical efficacy and safety of propiverine for treating patients with OAB have reported improvements in urinary frequency and incontinence, but not in urgency.

The aim of this study was to explore the efficacy of a daily regimen of propiverine at 20 mg (immediate release formulation) in improving urgency from baseline to 12 weeks of treatment in patients with OAB.

DETAILED DESCRIPTION:
12-week multi-center, prospective, parallel, double-blind, placebo-controlled trial

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Overactive bladder for at least 3 months
* 3 day- voiding diary

  * average urinary frequency ≥ 10 voids/24hrs
  * urgency ≥ 2 episodes/24hrs
* "moderate to severe" in the Indevus Urgency Severity Scale (IUSS)

Exclusion Criteria:

* clinically significant stress urinary incontinence
* polyuria of more than 3000 ml/24 hrs
* severe hepatic or renal diseases
* contraindications to the use of antimuscarinic drugs
* genitourinary conditions that could cause OAB symptoms such as urinary tract infection, genitourinary malignancy or interstitial cystitis
* uninvestigated hematuria
* clinically significant bladder outlet obstruction
* clinically significant pelvic organ prolapse
* being on a bladder-training program or having been on electrostimulation therapy two weeks before randomization or intention to start
* unstable dosages of drugs with anticholinergic side effects
* any other investigational drug taken up to 2 months prior to randomization
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Percent change in mean number of urgency episode | 12 weeks of treatment

SECONDARY OUTCOMES:
Change in the patients' perception of urgency | 12 weeks of treatment
Change in urgency severity/voids | 12 weeks of treatment
Change in sum of urgency severity/24 hours | 12 weeks of treatment
Changes in voiding frequency/24hrs, daytime and nocturnal voiding frequency/24 hours | 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Lee KS, Lee HW, Choo MS, Paick JS, Lee JG, Seo JT, Lee JZ, Lee YS, Yoon H, Park CH, Na YG, Jeong YB, Lee JB, Park WH. Urinary urgency outcomes after propiverine treatment for an overactive bladder: the 'Propiverine study on overactive bladder including urgency data'. BJU Int. 2010 Jun;105(11):1565-70. doi: 10.1111/j.1464-410X.2009.09050.x. Epub 2009 Nov 12. PMID 19912183